CLINICAL TRIAL: NCT02323581
Title: Feasibility, Safety, and Clinical Outcomes of Endovascular Treatment of Thoracoabdominal Aortic Aneurysms and Aortic Arch Aneurysms Using Fenestrated and Branched Stent Grafts
Brief Title: Endovascular Treatment of TAAA and Aortic Arch Aneurysms Using Fenestrated and Branched Stent Grafts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Darren Schneider, M.D. (Other)
Responsible Party: Sponsor-Investigator, Darren Schneider, M.D., Chief, Vascular Surgery and Endovascular Therapy, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 843522
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Aortic Aneurysm, Thoracoabdominal; Aortic Aneurysm, Thoracic; Aortic Dissection, Thoracoabdominal
Keywords: Thoracoabdominal; Aneurysm; Endovascular; Stent-Graft; Aortic Arch; BEVAR; FEVAR; Aorta; Aortic Dissection
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Aortic Aneurysm, Thoracic; Dissection, Abdominal Aorta; Aneurysm; Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- TAAA (thoracoabdominal aortic aneurysm) Study Arm (Experimental): Either the Off-the-Shelf TAAA device or the Physician-Specified TAAA Device will be implanted.
  The Off-the-Shelf TAAA Device is a standard configuration Zenith t-Branch with four branches for the mesenteric arteries and the renal arteries.
  The Physician-Specified TAAA Devices may include a combination of up to 5 fenestrations and branches for mesenteric and renal arteries. Branches will be used for downward-oriented mesenteric and renal arteries and fenestrations for renal arteries that project laterally or upwards.
  Interventions: Device: Endovascular treatment of Thoracoabdominal Aortic Aneurysm
- Aortic Arch Study Arm (Experimental): Physician-specified aortic arch stent graft device with up to 3 antegrade and/or retrograde branches or a physician-specified retrograde left subclavian branch stent-graft with double or triple wide scallop to the left common carotid artery] to treat aortic aneurysms involving the aortic arch in patients at high risk for open surgery.
  Interventions: Device: Endovascular treatment of Aortic Arch Aneurysms

INTERVENTIONS:
Device: Endovascular treatment of Thoracoabdominal Aortic Aneurysm — A TAAA is an abnormal enlargement (ballooning out) of the main artery (the aorta) and involves all or part of the aorta in your chest as well as all or part of the aorta in the abdomen. It also involves the part of the aorta where the arteries that bring blood to the liver, stomach and intestines and kidneys are attached.
  This investigational procedure that is being studied uses stent-grafts (cylindrical fabric tubes (grafts), with metal springs (stents) attached). The stent-grafts are placed inside the aneurysmal (weakened) area of the aorta to re-line it. These customized stent-grafts have special branches attached to them or openings (called "fenestrations") that are used to keep blood flowing to the arteries that supply the liver, stomach, intestines and kidneys. The investigational stent graft will be designed and custom-made specifically for your aneurysm.
  Arms: TAAA (thoracoabdominal aortic aneurysm) Study Arm
Device: Endovascular treatment of Aortic Arch Aneurysms — An aortic arch aneurysm is an abnormal enlargement (ballooning out) of the main artery (the aorta). The ascending aorta and aortic arch is the first part of the vessel as it exits the heart and makes a turn around the area of the collar bone. This part of the aorta gives branches that supply the head, brain and arms.
  The arch branch endovascular graft includes the main aortic arch portion and one to three cuffs (side branches) that allow the graft to be located in the aortic arch. The number of cuffs is decided based on the anatomy of your aneurysm. The arteries in the aortic arch are the innominate artery (Zone 0), left common carotid artery (Zone 1) and the left subclavian artery (Zone 2). These arteries supply the right arm and right side of the brain, the left side of the brain and the left arm, respectively.
  Arms: Aortic Arch Study Arm

SUMMARY:
Prospective, nonrandomized, single-center, two-arm study to assess the feasibility and safety and to evaluate clinical outcomes of endovascular repair of complex aortic aneurysms (thoracoabdominal aortic aneurysms and aortic arch aneurysms) in patients at high risk for open surgery.

DETAILED DESCRIPTION:
To assess the feasibility and safety and to evaluate clinical outcomes of endovascular repair of complex aortic aneurysms (thoracoabdominal aortic aneurysms and aortic arch aneurysms) in patients at high risk for open surgery in two study arms:

1. TAAA (thoracoabdominal aortic aneurysm) Study Arm: To assess the feasibility and safety and to evaluate clinical outcomes of endovascular stent graft implantation using either a multibranched stent graft (Off-the-Shelf TAAA Device) or custom-manufactured physician-specified branched and/or fenestrated stent graft (Physician-Specified TAAA Device) to treat aortic aneurysms involving the mesenteric and/or renal arteries (TAAA) in patients at high risk for open surgery.
2. Aortic Arch Study Arm: To assess the feasibility and safety and to evaluate clinical outcomes of endovascular stent graft implantation using 1) physician-specified aortic arch stent graft device with up to 3 antegrade and/or retrograde branches or 2) a physician-specified retrograde left subclavian branch stent-graft with double or triple wide scallop to the left common carotid artery] to treat aortic aneurysms involving the aortic arch in patients at high risk for open surgery.

ELIGIBILITY:
TAAA STUDY ARM

Inclusion Criteria:

1. Presence of TAAA in:

   1. Men with TAAA greater than or equal to 6 cm in diameter
   2. Women with TAAA greater than or equal to 5 cm in diameter
   3. Men with TAAA larger than 5 cm in diameter and enlarging at a rate of more than 10mm/year
   4. Women with TAAA larger than 4.5 cm in diameter and enlarging at a rate of more than 10mm/year or
   5. Men or women with TAAA and an iliac artery aneurysm greater than or equal to 4 cm in diameter
2. Life expectancy more than 2 years
3. Ability to give informed consent, complete pre-treatment assessments and comply with the follow-up schedule per protocol
4. Suitable arterial anatomy for endovascular TAAA repair with "TAAA device":

   1. Proximal aortic landing zone:

      * ≥ 20mm long
      * ≤ 40mm and ≥ 20mm diameter in parallel aorta
      * free from circumferential thrombus
      * ≤ 60 degrees angulation
   2. Mesenteric/renal aortic diameter ≥ 20mm
   3. Mesenteric arteries:

      * ≥ 10mm long segment of healthy artery for branch attachment
      * Diameter ≥ 4mm and ≤ 12mm
      * Absence of aberrant or early branching, aneurysm or dissection
   4. Renal arteries:

      * ≥ 10mm long segment of healthy artery for branch attachment
      * Diameter ≥ 4mm and ≤ 8mm
      * Absence of aberrant or early branching, aneurysm or dissection
   5. Iliac artery access:

      * ≥ 6mm diameter, and absence of severe calcification and tortuosity
      * Or, planned creation of surgical conduit for TAAA device delivery
   6. For patients with associated common iliac artery aneurysms (>20mm diameter), adequate internal and external iliac artery landing zones and common iliac artery luminal diameter (for iliac branch device use):

      * ≥ 10mm long segment of healthy internal iliac artery for branch attachment
      * Internal iliac diameter ≥ 5mm and ≤ 12mm
      * External iliac diameter ≥ 6mm diameter, and absence of severe calcification and tortuosity
      * Minimum common iliac artery luminal diameter ≥ 14mm
      * Or, in patients with bilateral common iliac artery aneurysms without suitable anatomy, planned surgical bypass to maintain patency of at least one internal iliac artery
5. Patients deemed high risk for open repair (meeting one, or more, of the following criteria):

   1. Age ≥ 65 year
   2. Cardiac disease:

      * CAD (history of MI or angina with positive stress test and not revascularizable)
      * LV Ejection fraction < 40%
      * Symptomatic CHF (NYHC Class II, III, or IV)
   3. Pulmonary disease:

      * Home oxygen therapy
      * FEV1 < 1.2 l/s
      * Vital capacity < 50% predicted
      * PaCO2 > 45 mm Hg or < 60 mm Hg
   4. Renal disease:

      * ESRD on dialysis
      * eGFR < 60
   5. Prior aortic surgery
   6. Hostile abdomen
   7. Portal hypertension (ascites or varices)
   8. Coagulopathy

AORTIC ARCH STUDY ARM

Inclusion Criteria:

1. Presence of aortic arch aneurysm in:

   1. Men with aortic arch aneurysm greater than or equal to 6 cm in diameter, or
   2. Women with aortic arch aneurysm greater than or equal to 5 cm in diameter, or
   3. Men with aortic arch aneurysm larger than 5 cm in diameter and enlarging at a rate of more than 10 mm/year, or
   4. Women with aortic arch aneurysm larger than 4.5 cm in diameter and enlarging at a rate of more than 10 mm/year, or
   5. Saccular aortic arch aneurysms deemed at significant risk for rupture based upon physician interpretation
2. Life expectancy more than 2 years
3. Ability to give informed consent, complete pre-treatment assessments and comply with the follow-up schedule per protocol.
4. Suitable arterial anatomy for endovascular aortic arch repair with "Aortic Arch Device":

   1. Aneurysm of the aortic arch beginning distal to the native coronary arteries or any patent coronary artery bypass
   2. Proximal aortic landing zone:

      * Native aorta or surgical graft
      * ≥ 20 mm long
      * ≤ 42 mm and ≥ 20 mm diameter in parallel aorta
      * free from circumferential thrombus
   3. Distal aortic landing zone:

      * Native aorta or surgical graft
      * ≥ 20 mm long
      * ≤ 42 mm and ≥ 20 mm diameter in parallel aorta
      * free from circumferential thrombus
      * ≥ 50mm length from native coronary arteries or patent coronary bypass graft to innominate artery
   4. Adequate supra-aortic trunk branch landing zone(s):

      * Innominate artery (if applicable):

        * Native vessel or surgical graft
        * Diameter: 8-22mm
        * Length of sealing zone ≥10mm
        * Acceptable tortuosity
        * Absence of dissection in landing zone
      * Left (or right) common carotid artery (if applicable):

        * Native vessel or surgical graft
        * Diameter 6-16mm
        * Length of sealing zone ≥10mm
        * Acceptable tortuosity
        * Absence of dissection in landing zone
      * Left (or right) subclavian artery (if applicable):

        * Native vessel or surgical graft
        * Diameter: 5-20mm
        * Length of sealing zone ≥10mm
        * Acceptable tortuosity
        * Absence of dissection in landing zone
   5. Iliac artery access:

      * ≥ 6mm diameter, and absence of severe calcification and tortuosity
      * Or, planned creation of surgical conduit for TAAA device delivery
5. Patients deemed high risk for open surgical aortic arch repair based upon consensus of both a qualified cardiac surgeon and a qualified vascular surgeon and meeting one, or more, of the following criteria):

   1. Age > 70 years-old
   2. Prior ascending or aortic arch repair
   3. Multiple (≥2) median sternotomies
   4. Ischemic cardiomyopathy with multi-level coronary artery disease and/or positive stress test
   5. Chronic pulmonary disease with FEV1 < 1500ml
   6. Chronic kidney disease with eGFR ≤ 60 ml/kg/hr
   7. Large aneurysm abutting the sternotomy
   8. Severe deconditioning or immobility
   9. Prior cervical irradiation
   10. Other medical condition associated with prohibitive high risk with open repair based upon multidisciplinary consensus (cardiac surgery and vascular surgery)

APPLIES TO BOTH STUDY ARMS

Exclusion Criteria:

1. Rupture, with hypotension (systolic bp < 90).
2. Pregnancy or breastfeeding.
3. Unwillingness or inability to comply with the follow up schedule.
4. Serious systemic or groin infection.
5. Uncorrectable coagulopathy.
6. Age < 18 years.
7. Mycotic aneurysm.
8. Known degenerative connective tissue disease, e.g., Marfan or Ehler-Danlos Syndrome (unless proximal implantation is into a previously placed surgical graft).
9. Known sensitivities or allergies to stainless steel, nitinol, polyester, solder (tin, silver), polypropylene, urethane or gold.
10. Participation in another in another investigational device or drug study within 1 year of treatment.
11. Unrelated concomitant major surgical or interventional procedure(s) within 30 days of treatment date (with the exception of staged procedures planned as part of treatment)
12. Body habitus that would inhibit X-ray visualization of the aorta.
13. Acute aortic dissection
14. Patients able and willing to be treated with a commercially available device or a device being evaluated in a manufacturer-sponsored pivotal study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Technical Success | Intraoperative
  Successful deployment of the TAAA device or Physician-Specified TAAA Devices, or Aortic Arch device & bridging covered stents into all targeted mesenteric & renal, or supra-aortic arteries with stent-graft & all branches patent by intraop angiography
Procedural Success | 30 days
  Technical success plus freedom from type I or III endoleak, loss of target vessel patency, death, major stroke, paralysis, new onset permanent hemodialysis, major amputation, & bowel infarction following deployment of the branched stent-graft.
Freedom from aneurysm-related mortality at 1 year | 1 year
  Survival from aneurysm-related death.
Treatment success at 12 months post-procedure | 1 year
  Composite endpoint which includes Technical Success, Procedural Success, and freedom from aneurysm-related mortality

SECONDARY OUTCOMES:
Target artery patency | Yearly through 5 years
  Imaging studies (CT Scans, Ultrasound and/or x-rays) are completed yearly to evaluate target artery patency.
Freedom from all-cause mortality | Yearly through 5 years
  Clinical evaluations are completed yearly and include bloodwork (WBC, Hemoglobin, Hematocrit, Platelets, BUN [Urea Nitrogen], Creatinine, eGFR), imaging scans (CT scans, Ultrasounds, and/or x-rays) and adverse event evaluation.
Freedom from reintervention | Yearly through 5 years
  Clinical evaluations are completed yearly and include bloodwork (WBC, Hemoglobin, Hematocrit, Platelets, BUN [Urea Nitrogen], Creatinine, eGFR), imaging scans (CT scans, Ultrasounds, and/or x-rays) and adverse event evaluation to determine if reintervention with the device is necessary.
Freedom from endoleak | Yearly through 5 years
  Imaging studies (CT Scans, Ultrasound and/or x-rays) are completed yearly to evaluate device integrity and any device leaks.
Freedom from aneurysm dilatation | Yearly through 5 years
  Imaging studies (CT Scans, Ultrasound and/or x-rays) are completed yearly to evaluate aneurysm size.
Freedom from serious adverse events (SAE) and major complications | Yearly through 5 years
  Clinical evaluations are completed yearly and include bloodwork (WBC, Hemoglobin, Hematocrit, Platelets, BUN [Urea Nitrogen], Creatinine, eGFR), imaging scans (CT scans, Ultrasounds, and/or x-rays) and adverse event evaluation.
Freedom from aneurysm rupture and conversion to open repair | Yearly through 5 years
  Clinical evaluations are completed yearly and include bloodwork (WBC, Hemoglobin, Hematocrit, Platelets, BUN [Urea Nitrogen], Creatinine, eGFR), imaging scans (CT scans, Ultrasounds, and/or x-rays) and adverse event evaluation to determine if aneurysm stability.
Freedom from stent graft migration and branch device migration | Yearly through 5 years
  Imaging studies (CT Scans, Ultrasound and/or x-rays) are completed yearly to evaluate device integrity and any device leaks.
Freedom from major stroke | Yearly through 5 years
  Clinical evaluations are completed yearly and include bloodwork (WBC, Hemoglobin, Hematocrit, Platelets, BUN [Urea Nitrogen], Creatinine, eGFR), imaging scans (CT scans, Ultrasounds, and/or x-rays) and adverse event evaluation.
Freedom from paralysis | Yearly through 5 years
  Clinical evaluations are completed yearly and include bloodwork (WBC, Hemoglobin, Hematocrit, Platelets, BUN [Urea Nitrogen], Creatinine, eGFR), imaging scans (CT scans, Ultrasounds, and/or x-rays) and adverse event evaluation.
Freedom from onset permanent hemodialysis | Yearly through 5 years
  Clinical evaluations are completed yearly and include bloodwork (WBC, Hemoglobin, Hematocrit, Platelets, BUN [Urea Nitrogen], Creatinine, eGFR), imaging scans (CT scans, Ultrasounds, and/or x-rays) and adverse event evaluation.
Freedom from amputation | Yearly through 5 years
  Clinical evaluations are completed yearly and include bloodwork (WBC, Hemoglobin, Hematocrit, Platelets, BUN [Urea Nitrogen], Creatinine, eGFR), imaging scans (CT scans, Ultrasounds, and/or x-rays) and adverse event evaluation.
Freedom from bowel infarction | Yearly through 5 years
  Clinical evaluations are completed yearly and include bloodwork (WBC, Hemoglobin, Hematocrit, Platelets, BUN [Urea Nitrogen], Creatinine, eGFR), imaging scans (CT scans, Ultrasounds, and/or x-rays) and adverse event evaluation.
Freedom from loss of target vessel patency | Yearly through 5 years
  Imaging studies (CT Scans, Ultrasound and/or x-rays) are completed yearly to evaluate device integrity and any device leaks.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Schneider, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - New York Presbyterian Hospital, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Meltzer AJ, Connolly PH, Ellozy S, Schneider DB. Patient-reported Quality of Life after Endovascular Repair of Thoracoabdominal Aortic Aneurysms. Ann Vasc Surg. 2017 Oct;44:164-170. doi: 10.1016/j.avsg.2017.04.009. Epub 2017 May 17. PMID 28527678
- [Background] Stern JR, Ellozy SH, Connolly PH, Meltzer AJ, Schneider DB. Utility and safety of axillary conduits during endovascular repair of thoracoabdominal aneurysms. J Vasc Surg. 2017 Sep;66(3):705-710. doi: 10.1016/j.jvs.2016.12.107. Epub 2017 Mar 1. PMID 28259569
- [Background] Schneider DB, Agrusa CJ, Ellozy SH, Connolly PH, Meltzer AJ, Graham AR, Michelassi F. Analysis of the Learning Curve and Patient Outcomes of Endovascular Repair of Thoracoabdominal Aortic Aneurysms Using Fenestrated and Branched Stent Grafts: Prospective, Nonrandomized, Single-center Physician-sponsored Investigational Device Exemption Clinical Study. Ann Surg. 2018 Oct;268(4):640-649. doi: 10.1097/SLA.0000000000002960. PMID 30080733
- [Background] Dias-Neto M, Vacirca A, Huang Y, Baghbani-Oskouei A, Jakimowicz T, Mendes BC, Kolbel T, Sobocinski J, Bertoglio L, Mees B, Gargiulo M, Dias N, Schanzer A, Gasper W, Beck AW, Farber MA, Mani K, Timaran C, Schneider DB, Pedro LM, Tsilimparis N, Haulon S, Sweet MP, Ferreira E, Eagleton M, Yeung KK, Khashram M, Jama K, Panuccio G, Rohlffs F, Mesnard T, Chiesa R, Kahlberg A, Schurink GW, Lemmens C, Gallitto E, Faggioli G, Karelis A, Parodi E, Gomes V, Wanhainen A, Habib M, Colon JP, Pavarino F, Baig MS, Gouveia E Melo REC, Crawford S, Zettervall SL, Garcia R, Ribeiro T, Alves G, Goncalves FB, Kappe KO, Mariko van Knippenberg SE, Tran BL, Gormley S, Oderich GS; International Multicenter Aortic Research Group. Outcomes of Elective and Non-elective Fenestrated-branched Endovascular Aortic Repair for Treatment of Thoracoabdominal Aortic Aneurysms. Ann Surg. 2023 Oct 1;278(4):568-577. doi: 10.1097/SLA.0000000000005986. Epub 2023 Jul 3. PMID 37395613
- [Background] Finnesgard EJ, Beck AW, Eagleton MJ, Farber MA, Gasper WJ, Lee WA, Oderich GS, Schneider DB, Sweet MP, Timaran CH, Simons JP, Schanzer A; United States Aortic Research Consortium. Severity of acute kidney injury is associated with decreased survival after fenestrated and branched endovascular aortic aneurysm repair. J Vasc Surg. 2023 Oct;78(4):892-901. doi: 10.1016/j.jvs.2023.05.034. Epub 2023 Jun 16. PMID 37330702
- [Background] Abdelhalim MA, Tenorio ER, Oderich GS, Haulon S, Warren G, Adam D, Claridge M, Butt T, Abisi S, Dias NV, Kolbel T, Gallitto E, Gargiulo M, Gkoutzios P, Panuccio G, Kuzniar M, Mani K, Mees BM, Schurink GW, Sonesson B, Spath P, Wanhainen A, Schanzer A, Beck AW, Schneider DB, Timaran CH, Eagleton M, Farber MA, Modarai B; Multicenter International Aortic Research Group. Multicenter trans-Atlantic experience with fenestrated-branched endovascular aortic repair of chronic post-dissection thoracoabdominal aortic aneurysms. J Vasc Surg. 2023 Oct;78(4):854-862.e1. doi: 10.1016/j.jvs.2023.05.053. Epub 2023 Jun 13. PMID 37321524
- [Background] Aucoin VJ, Motyl CM, Novak Z, Eagleton MJ, Farber MA, Gasper W, Oderich GS, Mendes B, Schanzer A, Tenorio E, Timaran CH, Schneider DB, Sweet MP, Zettervall SL, Beck AW; U.S. Aortic Research Consortium. Predictors and outcomes of spinal cord injury following complex branched/fenestrated endovascular aortic repair in the US Aortic Research Consortium. J Vasc Surg. 2023 Jun;77(6):1578-1587. doi: 10.1016/j.jvs.2023.01.205. Epub 2023 Apr 13. PMID 37059239
- [Background] Tenorio ER, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Parodi FE, Gasper WJ, Beck AW, Sweet MP, Huang Y, Oderich GS; U.S. Fenestrated and Branched Aortic Research Consortium. Mid-term Renal and Mesenteric Artery Outcomes During Fenestrated and Branched Endovascular Aortic Repair for Complex Abdominal and Thoracoabdominal Aortic Aneurysms in the United States Aortic Research Consortium. Ann Surg. 2023 Oct 1;278(4):e893-e902. doi: 10.1097/SLA.0000000000005859. Epub 2023 Apr 13. PMID 37051912
- [Background] Tenorio ER, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Parodi FE, Gasper WJ, Beck AW, Sweet MP, Zettervall SL, Huang Y, Oderich GS; U.S. Fenestrated and Branched Aortic Research Consortium. Effect of bridging stent graft selection for directional branches on target artery outcomes of fenestrated-branched endovascular aortic repair in the United States Aortic Research Consortium. J Vasc Surg. 2023 Jul;78(1):10-28.e3. doi: 10.1016/j.jvs.2023.03.025. Epub 2023 Mar 21. PMID 36948277
- [Background] Heslin RT, Blakeslee-Carter J, Novak Z, Eagleton MJ, Farber MA, Oderich GS, Schanzer A, Timaran CH, Schneider DB, Sweet MP, Beck AW. Aneurysm extent-based mortality differences in complex endovascular repair of thoracoabdominal aneurysms in the Vascular Quality Initiative and the United States Aortic Research Consortium. J Vasc Surg. 2023 Jul;78(1):1-9.e3. doi: 10.1016/j.jvs.2023.02.020. Epub 2023 Mar 14. PMID 36921644
- [Background] Dias-Neto M, Tenorio ER, Huang Y, Jakimowicz T, Mendes BC, Kolbel T, Sobocinski J, Bertoglio L, Mees B, Gargiulo M, Dias N, Schanzer A, Gasper W, Beck AW, Farber MA, Mani K, Timaran C, Schneider DB, Pedro LM, Tsilimparis N, Haulon S, Sweet M, Ferreira E, Eagleton M, Yeung KK, Khashram M, Vacirca A, Lima GB, Baghbani-Oskouei A, Jama K, Panuccio G, Rohlffs F, Chiesa R, Schurink GW, Lemmens C, Gallitto E, Faggioli G, Karelis A, Parodi E, Gomes V, Wanhainen A, Dean A, Colon JP, Pavarino F, E Melo RG, Crawford S, Garcia R, Ribeiro T, Kappe KO, van Knippenberg SEM, Tran BL, Gormley S, Oderich GS; International Aortic Research Consortium. Comparison of single- and multistage strategies during fenestrated-branched endovascular aortic repair of thoracoabdominal aortic aneurysms. J Vasc Surg. 2023 Jun;77(6):1588-1597.e4. doi: 10.1016/j.jvs.2023.01.188. Epub 2023 Jan 31. PMID 36731757
- [Background] Chamseddin K, Timaran CH, Oderich GS, Tenorio ER, Farber MA, Parodi FE, Schneider DB, Schanzer A, Beck AW, Sweet MP, Zettervall SL, Mendes B, Eagleton MJ, Gasper WJ; U.S. Aortic Research Consortium. Comparison of upper extremity and transfemoral access for fenestrated-branched endovascular aortic repair. J Vasc Surg. 2023 Mar;77(3):704-711. doi: 10.1016/j.jvs.2022.10.009. Epub 2022 Oct 17. PMID 36257344
- [Background] Zettervall SL, Tenorio ER, Schanzer A, Oderich GS, Timaran CH, Schneider DB, Eagleton M, Farber MA, Gasper WJ, Beck AW, Sweet MP; U.S. Fenestrated and Branched Aortic Research Consortium. Secondary interventions after fenestrated/branched aneurysm repairs are common and nondetrimental to long-term survival. J Vasc Surg. 2022 May;75(5):1530-1538.e4. doi: 10.1016/j.jvs.2021.11.074. Epub 2021 Dec 23. PMID 34954272
- [Background] Edman NI, Schanzer A, Crawford A, Oderich GS, Farber MA, Schneider DB, Timaran CH, Beck AW, Eagleton M, Sweet MP; U.S. Fenestrated and Branched Aortic Research Consortium. Sex-related outcomes after fenestrated-branched endovascular aneurysm repair for thoracoabdominal aortic aneurysms in the U.S. Fenestrated and Branched Aortic Research Consortium. J Vasc Surg. 2021 Sep;74(3):861-870. doi: 10.1016/j.jvs.2021.02.046. Epub 2021 Mar 26. PMID 33775747
- [Background] Timaran CH, Oderich GS, Tenorio ER, Farber MA, Schneider DB, Schanzer A, Beck AW, Sweet MP; Aortic Research Consortium. Expanded Use of Preloaded Branched and Fenestrated Endografts for Endovascular Repair of Complex Aortic Aneurysms. Eur J Vasc Endovasc Surg. 2021 Feb;61(2):219-226. doi: 10.1016/j.ejvs.2020.11.001. Epub 2020 Nov 28. PMID 33262091
- [Background] Banga P, Oderich GS, Farber M, Reis de Souza L, Tenorio ER, Timaran C, Schneider DB, Baumgardt Barbosa Lima G, Barreira Marcondes G, Timaran D. Impact of Number of Vessels Targeted on Outcomes of Fenestrated-Branched Endovascular Repair for Complex Abdominal Aortic Aneurysms. Ann Vasc Surg. 2021 Apr;72:98-105. doi: 10.1016/j.avsg.2020.09.063. Epub 2020 Nov 21. PMID 33227467
- [Background] Aucoin VJ, Eagleton MJ, Farber MA, Oderich GS, Schanzer A, Timaran CH, Schneider DB, Sweet MP, Beck AW. Spinal cord protection practices used during endovascular repair of complex aortic aneurysms by the U.S. Aortic Research Consortium. J Vasc Surg. 2021 Jan;73(1):323-330. doi: 10.1016/j.jvs.2020.07.107. Epub 2020 Aug 31. PMID 32882346
- [Background] Kitpanit N, Ellozy SH, Connolly PH, Agrusa CJ, Lichtman AD, Schneider DB. Risk factors for spinal cord injury and complications of cerebrospinal fluid drainage in patients undergoing fenestrated and branched endovascular aneurysm repair. J Vasc Surg. 2021 Feb;73(2):399-409.e1. doi: 10.1016/j.jvs.2020.05.070. Epub 2020 Jul 5. PMID 32640318
- [Background] Tenorio ER, Oderich GS, Farber MA, Schneider DB, Timaran CH, Schanzer A, Beck AW, Motta F, Sweet MP; U.S. Fenestrated and Branched Aortic Research Consortium Investigators. Outcomes of endovascular repair of chronic postdissection compared with degenerative thoracoabdominal aortic aneurysms using fenestrated-branched stent grafts. J Vasc Surg. 2020 Sep;72(3):822-836.e9. doi: 10.1016/j.jvs.2019.10.091. Epub 2019 Dec 25. PMID 31882309
- [Background] Agrusa CJ, Connolly PH, Ellozy SH, Schneider DB. Safety and Effectiveness of Percutaneous Axillary Artery Access for Complex Aortic Interventions. Ann Vasc Surg. 2019 Nov;61:326-333. doi: 10.1016/j.avsg.2019.05.046. Epub 2019 Aug 5. PMID 31394224
- [Background] Banks CA, Novak Z, Spangler EL, Schanzer A, Farber MA, Sweet MP, Oderich G, Timaran CH, Lee A, Schneider DB, Eagleton MJ, Gasper W, Beck AW. Preoperative risk factors for 1-year mortality in patients undergoing fenestrated endovascular aortic aneurysm repair in the US Aortic Research Consortium. J Vasc Surg. 2024 Sep;80(3):724-735.e3. doi: 10.1016/j.jvs.2024.04.063. Epub 2024 May 6. PMID 38718849
- [Background] Blakeslee-Carter J, Novak Z, Jansen JO, Schanzer A, Eagleton MJ, Farber MA, Gasper W, Lee WA, Oderich GS, Timaran CH, Schneider DB, Sweet MP, Beck AW. Prospective randomized pilot trial comparing prophylactic and therapeutic cerebrospinal fluid drainage during complex endovascular thoracoabdominal aortic aneurysm repair. J Vasc Surg. 2024 Jul;80(1):11-19. doi: 10.1016/j.jvs.2024.02.041. Epub 2024 Apr 6. PMID 38614137
- [Background] Fan EY, Schanzer A, Beck AW, Eagleton MJ, Farber MA, Gasper WJ, Lee WA, Oderich GS, Parodi FE, Schneider DB, Sweet MP, Timaran CH, Simons JP; US Aortic Research Consortium. Practice patterns of antiplatelet and anticoagulant therapy after fenestrated/branched endovascular aortic repair. J Vasc Surg. 2024 Oct;80(4):968-978.e3. doi: 10.1016/j.jvs.2024.05.041. Epub 2024 May 23. PMID 38796031
- [Background] Oderich GS, Huang Y, Harmsen WS, Tenorio ER, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Gasper WJ, Beck AW, Sweet MP, Lee WA; United States Aortic Research Consortium. Early and Late Aortic-Related Mortality and Rupture After Fenestrated-Branched Endovascular Aortic Repair of Thoracoabdominal Aortic Aneurysms: A Prospective Multicenter Cohort Study. Circulation. 2024 Oct 22;150(17):1343-1353. doi: 10.1161/CIRCULATIONAHA.123.068234. Epub 2024 Jul 11. PMID 38989575
- [Background] Al Adas Z, Uceda D, Mazur A, Zehner K, Agrusa CJ, Wang G, Schneider DB. Safety and learning curve of percutaneous axillary artery access for complex endovascular aortic procedures. J Vasc Surg. 2024 Mar;79(3):487-496. doi: 10.1016/j.jvs.2023.10.048. Epub 2023 Oct 31. PMID 37918698
- [Derived] Mesnard T, Huang Y, Schanzer A, Timaran CH, Schneider DB, Mendes BC, Eagleton MJ, Farber MA, Parodi FE, Gasper WJ, Beck AW, Sweet MP, Zetterval SL, Lee A, Oderich GS; United States Aortic Research Consortium. Multicenter Prospective Evaluation of Patient Radiation Exposure During Fenestrated-Branched Endovascular Aortic Repair: A Ten-year Experience. Ann Surg. 2025 Feb 18. doi: 10.1097/SLA.0000000000006676. Online ahead of print. PMID 39963789